CLINICAL TRIAL: NCT04600011
Title: A Novel Tele-Neurorehabilitation Program Aimed at Reducing Fall Risk in Parkinson's Disease Patients
Brief Title: Telerehabilitation for Parkinson's Disease
Acronym: TelerehabPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Mitra Afshari, Assistant Professor of Neurological Sciences, Rush University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19050804-IRB01
Record Dates: First submitted 2020-02-07; First posted 2020-10-23 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease; Telemedicine
MeSH Terms: conditions — Parkinson Disease | interventions — Restraint, Physical; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Pilot feasibility study, non-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TELEREHABILITATION ARM (Other): ARM 1: The TELEREHABILITATION ARM where participants receive the full originally-intended protocol that includes one initial in-person PT/OT evaluation, four virtual PT/OT visits, and one final in-person (or virtual, if in-person is not possible) PT/OT evaluation. The study duration for Arm 1 is about 10 weeks of the primary intervention as described with 3- and 6-month follow-up calls. The mobile virtual platform for Arm 1 is comprised of a tablet on a height-adjustable rotating tablet floor stand with a gooseneck and wheels.
  Interventions: Other: Physical and occupational therapy (PT/OT)
- VIRTUAL HOME SAFETY EVALUATIONS (HSE)-ONLY ARM (Other): ARM 2: The VIRTUAL HOME SAFETY EVALUTIONS (HSE)-ONLY ARM where participants ONLY receive the virtual home safety evaluations and surveillance that are built into the original protocol of three of the four tele-OT visits that is being used in Arm 1. The study duration for Arm 2 is about 6 weeks of the primary intervention as described with 3-month and 6-month follow-up calls. The mobile virtual platform for Arm 2 is comprised of a tablet OR smartphone that will be guided through the home by the care partner only and not the patient.
  Interventions: Other: Home Safety Evaluation (HSE)

INTERVENTIONS:
Other: Physical and occupational therapy (PT/OT) — Neurologic-specialized and -certified physical and occupational therapists will provide each participant with an initial in-person PT/OT evaluation/treatment session with oversight from a Movement Disorders Neurologist, followed by 4 "virtual home visits" with tele-PT/OT and care partner supervision every 2 weeks, and culminating with a final in-person evaluation, all with a focus on personalized training in core areas contributing to a patient's individual fall risk, much like in-person visits. Virtual home safety surveillance with the mobile virtual platform is an additional feature of this intervention that aims to optimize the home environment to reduce external factors contributing to fall risk.
  Arms: TELEREHABILITATION ARM
Other: Home Safety Evaluation (HSE) — The VIRTUAL HOME SAFETY EVALUTIONS (HSE)-ONLY ARM where participants ONLY receive the virtual home safety evaluations and surveillance that are built into the original protocol of three of the four tele-OT visits that is being used in Arm 1. The study duration for Arm 2 is about 6 weeks of the primary intervention as described with 3-month and 6-month follow-up calls. The mobile virtual platform for Arm 2 is comprised of a tablet OR smartphone that will be guided through the home by the care partner only and not the patient.
  Arms: VIRTUAL HOME SAFETY EVALUATIONS (HSE)-ONLY ARM

SUMMARY:
Our primary objective in this 10-week pilot study is to demonstrate the feasibility of using videoconferencing technology to provide Parkinson's Disease (PD) patients, alongside their supervising care partners, specialized physical and occupational therapy (PT/OT) focused on neurorehabilitation that ultimately aims to reduce fall risk. This therapy is similar to what a PD patient could receive in-person with neurologic-certified physical therapists and occupational therapists with significant experience working with PD patients and addressing their needs, but it is delivered through a virtual platform. Feasibility is defined by measures of adherence, retention, and safety.

The specialized PT and OT measurement tools and strategies used in this study are in-line with the most current formal evidence-based guidelines/recommendations available for therapy in PD: European Physiotherapy Guideline for Parkinson's Disease, Parkinson Evidence Database to Guide Effectiveness (PD-EDGE) Task Force and Guidelines for Occupational Therapy in Parkinson's Disease Rehabilitation.

The study duration is approximately 10 weeks of the primary telerehabilitation intervention and a 2 follow-up phone calls at the 3- and 6-month timepoints. There will be one baseline in-person evaluation and one final in-person evaluation following the completion of all televisits. The enrollment target is up to 15-20 patient and care partner (P+CP) pairs, meaning 30-40 subjects total. There are no controls for this study.

DETAILED DESCRIPTION:
Gait dysfunction, postural instability, and freezing-of-gait (FOG) ultimately develop in about 80% of PD patients, which lead to falls and advancing disability. This is significant because the consequences of falls are far-reaching: accelerating immobility due to heightened fear-of-falling, reducing quality of life and independence, and increasing healthcare utilization and costs. Thus, there is an urgent need to expand evidence- based outpatient neurologic-PT/OT services to community-dwelling PD patients to reduce fall risk.

This research proposal will address this unmet need by determining whether tele-neurorehabilitation is a care model that can be executed safety for PD patients to provide these services from well-trained therapists who are not easily accessible otherwise. This feasibility data is critical in the development of a novel tele-neurorehabilitation protocol and randomized-controlled efficacy trial thereafter.

The impact of the intended research is to demonstrate the feasibility and preliminary efficacy of this novel teleconferencing-based delivery of gait and balance exercises/strategies with guided instruction much like one would receive in-person but in the comfort of one's own home. By demonstrating the feasibility and preliminary efficacy of this pilot program, subsequent long-term goals are to apply for larger sources of funding to sustain the program. By leveraging the data gained from these studies it is anticipated the practice of telerehabilitation will be expanded and improved; and ultimately its efficacy to health care policy providers and insurers for potential reimbursement will be demonstrated.

The researchers intend to enroll 15-20 individuals with mild-moderate PD into our proposed novel telerehabilitation program, where patients will receive tele-PT/OT home visits and home-safety surveillance with neurologic-specialized therapists who are experienced with the core problem areas seen in PD patients. The intended clinical impact is to improve gait/balance function and postural stability, and thus reduce falls in patients with PD. With the remote telecommunications intervention, we aim to enable the additional clinical impact of expanding access to therapy for people with PD that otherwise would have significant difficulty obtaining this type of multiple-visit, individually-tailored, and specialized therapy care due to travel burden and cost.

ELIGIBILITY:
Subject Inclusion Criteria:

1. Subject's age is greater than or equal to 18.
2. Subject has a diagnosis of Idiopathic Parkinson's Disease according to established criteria and this has been confirmed by a Movement Disorders Neurologist.
3. Subject's Movement Disorders Neurologist believes he/she would benefit from specialized physical and occupational therapy to reduce fall risk.
4. Subject's Idiopathic Parkinson's Disease is Hoehn and Yahr stage 2 or 3 in the "OFF"-medication state (stage 2 defined by bilateral or midline symptoms with less than or equal to 2 steps back on the pull test with self-recovery; stage 3 is defined by more than 2 steps back on the pull test with or without self-recovery, or no steps back and requiring assistance to recover).
5. Subject demonstrates the ability to utilize the virtual platform at their initial in-person evaluation.
6. Subject has been on a stable medication regimen for the treatment of Idiopathic Parkinson's Disease for the month preceding the baseline in-person visit, and has the ability to maintain stable dosing for the duration of the 10-week primary intervention.
7. Subject has home Wi-Fi access for the tele-neurorehabilitation home visits and a personal tablet with Wi-Fi connectivity.

Care Partner Inclusion Criteria:

1. Care partner's age is greater than or equal to 18.
2. Care partner has been the primary caregiver for >6 months and will remain so for at least 10 weeks to the study subject.
3. Care partner has the ability and desire to participate in all of the study visits with the study subject, including the tele-neurorehabilitation home visits.
4. Care partner has the ability and desire to provide stand-by assistance, but in the setting of a gait belt, to the study subject during tele-neurorehabilitation home visits.

Subject Exclusion Criteria:

1. Subject is non-English speaking.
2. Subject has only a provisional diagnosis of Idiopathic Parkinson's Disease or atypical features suggestive of an alternative diagnosis.
3. Subject has and additional significant neurologic diagnosis that may render him/her with neurologic deficits that may affect gait and balance.
4. Subject has another destabilizing chronic medical condition which may warrant frequent hospitalization or render the patient unable to participate in physical activity.
5. Subject requires more than just stand-by assistance for gait and balance.
6. Subject is reliant on mobility devices to walk (walkers, cane, walking sticks, motorized scooter, etc).
7. Subject is receiving physical therapy elsewhere during the month preceding the study and during the duration of the study.
8. Subject has no care partner available to participate in all of the study visits.
9. Subject is unable to follow direction or consent to research.
10. Subject is unable to commit to the study-related activities and/or schedule of events.

Care Partner Exclusion Criteria:

1. Care partner is non-English speaking.
2. Care partner is unable to follow direction or consent to research.
3. Care partner is unable to commit to the study-related activities and/or schedule of events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Adherence Measure - 1: | Through study completion of approximately 18 months.
  (1) The proportion of scheduled protocol-driven tele-PT and tele-OT visits that were completed.
Adherence Measure - 2: | Through study completion of approximately 18 months.
  (2) The proportion of scheduled protocol-driven PT/OT exercises/activities that could be completed virtually as assessed by the instructing study therapist.
Adherence Measure - 3: | Through study completion of approximately 18 months.
  (3) Qualitative categorization of limitations in performing tele-PT and tele-OT visits and PT/OT exercises/activities virtually into patient-related, technology-related, or environmentally-related limitations
Retention Measures: | Through study completion of approximately 18 months.
  The proportion of patient and care partner (P+CP) pairs that enrolled and were able to complete the study, i.e. study drop-out rate.
Safety Measures: | Through study completion of approximately 18 months.
  The number and nature of adverse and serious adverse events that occurred due to participation in the study, and the proportion deemed a result of study-related interventions.

SECONDARY OUTCOMES:
Goals Attainment Scale Score: | Through study completion of approximately 18 months.
  Change in Goals Attainment Scale score (GAS) from baseline across the 10-week program and at the 3- and 6-month follow-ups (Visits 1, 3, 5, 6, Follow-up Call 1-2) for 3 patient-specific PT goals under the following categories: gait/balance, strengthening, and physical endurance, and 2 patient-specific OT goals under the category of activities-of-daily-living/home safety, defined at the baseline assessment.
Falls Diary; | Through study completion of approximately 18 months.
  The change in falls frequency using the Falls Diary from baseline across the 10-week program and at the 3- and 6-month follow-ups (Visits 1, 3, 5, 6, Follow-up Call 1-2).
Activities-Specific Balance Scale: | Through study completion of approximately 18 months.
  The change in gait confidence from baseline using the Activities-Specific Balance Confidence scale (ABC scale) across the 10-week program and at the 3- and 6-month follow-ups (Visits 1, 2-6, Follow-Up Call 1-2)
Five-Times Sit-to-Stand Test: | Through study completion of approximately 18 months.
  The change in postural stability from baseline using the Five-Times Sit-to-Stand test (FTSTS) across the 10-week program to be performed both in-person and virtually (Visits 1, 3, 5, 6).
In-Person Objective Therapy Measure - 1: | Through study completion of approximately 18 months.
  The change in the following in-person assessment Mini-Balance Evaluation Systems Test (mini-BESTest) from baseline to post-intervention (Visits 1 and 6).
In-Person Objective Therapy Measure - 2: | Through study completion of approximately 18 months.
  The change in the following in-person assessment Rapid Turns Test (RTT) from baseline to post-intervention (Visits 1 and 6).
In-Person Objective Therapy Measure - 3: | Through study completion of approximately 18 months.
  The change in the following in-person assessment Timed Up and Go (TUG)from baseline to post-intervention (Visits 1 and 6).
In-Person Objective Therapy Measures - 4: | Through study completion of approximately 18 months.
  The change in the following in-person assessment Timed Up and Go-Cognitive (TUG-Cognitive) from baseline to post-intervention (Visits 1 and 6).
In-Person Objective Therapy Measure - 5: | Through study completion of approximately 18 months.
  The change in the following in-person assessment 10-Meter Walk Time (10MWT) from baseline to post-intervention (Visits 1 and 6).
In-Person Objective Therapy Measures - 6: | Through study completion of approximately 18 months.
  The change in the following in-person assessment 2-Minute Walk Distance Test (2MWT) from baseline to post-intervention (Visits 1 and 6).
Rapid Turns Test: | Through study completion of approximately 18 months.
  The change in freezing-of-gait from baseline using the Rapid Turns Test (RTT) across the 10-week program to be performed both in-person and virtually (Visits 1, 3, 5, and 6).
Parkinson's Disease Questionnaire-39: | Through study completion of approximately 18 months.
  The change in quality-of-life (QOL) using the Parkinson's Disease Questionnaire-39 (PDQ-39) from baseline to post-intervention (Visits 1 and 6).
Home Exercise Program: | Through study completion of approximately 18 months.
  The proportion of patients who were able to adhere to their recommended home exercise program (HEP) in between study visits as assessed by weekly coordinator phone calls.

OTHER OUTCOMES:
APDM Mobility Lab Sensor Data: | Through study completion of approximately 18 months.
  Change in measures of comprehensive gait, functional mobility, and postural sway analyses from baseline (Visit 1) to post-intervention (Visit 6) using the APDM Mobility LabTM six-inertial sensory system (APDMTM, Oregon) in the "OFF" medication state in a subset of 5-10 patients.
"Telehealth Satisfaction Survey": | Through study completion of approximately 18 months.
  Qualitative assessment using Likert-based questions and qualitative assessment of the patient, care partner, and study therapists' satisfaction with and perspectives on tele-neurorehabilitation virtual home visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mitra Afshari, MD, MPH, Principal Investigator — Rush University
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marras C, Beck JC, Bower JH, Roberts E, Ritz B, Ross GW, Abbott RD, Savica R, Van Den Eeden SK, Willis AW, Tanner CM; Parkinson's Foundation P4 Group. Prevalence of Parkinson's disease across North America. NPJ Parkinsons Dis. 2018 Jul 10;4:21. doi: 10.1038/s41531-018-0058-0. eCollection 2018. PMID 30003140
- [Background] Macht M, Kaussner Y, Moller JC, Stiasny-Kolster K, Eggert KM, Kruger HP, Ellgring H. Predictors of freezing in Parkinson's disease: a survey of 6,620 patients. Mov Disord. 2007 May 15;22(7):953-6. doi: 10.1002/mds.21458. PMID 17377927
- [Background] Hely MA, Morris JG, Reid WG, Trafficante R. Sydney Multicenter Study of Parkinson's disease: non-L-dopa-responsive problems dominate at 15 years. Mov Disord. 2005 Feb;20(2):190-9. doi: 10.1002/mds.20324. PMID 15551331
- [Background] Poewe W. The natural history of Parkinson's disease. J Neurol. 2006 Dec;253 Suppl 7:VII2-6. doi: 10.1007/s00415-006-7002-7. PMID 17131223
- [Background] Low V, Ben-Shlomo Y, Coward E, Fletcher S, Walker R, Clarke CE. Measuring the burden and mortality of hospitalisation in Parkinson's disease: A cross-sectional analysis of the English Hospital Episodes Statistics database 2009-2013. Parkinsonism Relat Disord. 2015 May;21(5):449-54. doi: 10.1016/j.parkreldis.2015.01.017. Epub 2015 Feb 17. PMID 25737205
- [Background] Wielinski CL, Erickson-Davis C, Wichmann R, Walde-Douglas M, Parashos SA. Falls and injuries resulting from falls among patients with Parkinson's disease and other parkinsonian syndromes. Mov Disord. 2005 Apr;20(4):410-415. doi: 10.1002/mds.20347. PMID 15580552
- [Background] Pressley JC, Louis ED, Tang MX, Cote L, Cohen PD, Glied S, Mayeux R. The impact of comorbid disease and injuries on resource use and expenditures in parkinsonism. Neurology. 2003 Jan 14;60(1):87-93. doi: 10.1212/wnl.60.1.87. PMID 12525724
- [Derived] Afshari M, Hernandez AV, Joyce JM, Hauptschein AW, Trenkle KL, Stebbins GT, Goetz CG. A Novel Home-Based Telerehabilitation Program Targeting Fall Prevention in Parkinson Disease: A Preliminary Trial. Neurol Clin Pract. 2024 Feb;14(1):e200246. doi: 10.1212/CPJ.0000000000200246. Epub 2024 Jan 5. PMID 38213401

DOCUMENTS (1):
  • Informed Consent Form (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT04600011/ICF_000.pdf